CLINICAL TRIAL: NCT06270238
Title: Efficacy of Personalized Repetitive Transcranial Magnetic Stimulation Protocol Based on Functional Reserve to Enhance Upper Limb Function in Subacute Stroke Patients: A Multi Center, Randomized, Single Blind, Parallel Group Prospective Clinical Trial
Brief Title: Efficacy of Personalized Repetitive Transcranial Magnetic Stimulation Protocol Based on Functional Reserve to Enhance Upper Limb Function in Subacute Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: National Research Foundation of Korea (Other); Ministry of Food and Drug Safety, Korea (Other Government); Seoul National University Hospital (Other); Bucheon St. Mary's Hospital (Other); Saint Vincent's Hospital, Korea (Other); Severance Hospital (Other); Kumoh National Institute of Technology (Unknown); NEUROPHET (Industry)
Responsible Party: Principal Investigator, Won Hyuk Chang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-11-164
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Stroke; rTMS; Functional reserve
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: prospective, single-blind with blind observer, parallel-group design, multi-center, randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, assessors, and investigators will be blinded, not be aware of the group allocation. Statistical analysis will also be conducted by data analysts without awareness of the group allocation. Only clinicians applying rTMS intervention will not be blinded, as they will apply rTMS over different stimulation sites based on the protocols. Blinding will be continued until the end of the study, including data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High-Frequency1 (Experimental): Confirmed responses in TMS-induced MEP: Preserved ipsilateral corticospinal tract.
  High-frequency rTMS over ipsilateral primary motor cortex will be applied.
  Interventions: Device: High-Frequency1
- cTBS1 (Active Comparator): Confirmed responses in TMS-induced MEP: Preserved ipsilateral corticospinal tract.
  continous Theta Burst Stimulation (cTBS) protocol of rTMS over contralateral primary motor cortex will be applied.
  Interventions: Device: cTBS1
- High-Frequency2 (Experimental): Absent responses in TMS-induced MEPs, but confirmed corticospinal tract integrity in DTI; Preserved ipsilateral alternative corticospinal tract.
  High-frequency rTMS over ipsilateral premotor cortex will be applied.
  Interventions: Device: High-Frequency2
- cTBS2 (Active Comparator): Absent responses in TMS-induced MEPs, but confirmed corticospinal tract integrity in DTI; Preserved ipsilateral alternative corticospinal tract.
  continous Theta Burst Stimulation (cTBS) protocol of rTMS over contralateral primary motor cortex will be applied.
  Interventions: Device: cTBS2
- High-Frequency3 (Experimental): Absent responses in all ipsilateral corticospinal tract.
  High-frequency rTMS over contralateral primary motor cortex will be applied.
  Interventions: Device: High-Frequency3
- cTBS3 (Active Comparator): Absent responses in all ipsilateral corticospinal tract.
  continous Theta Burst Stimulation (cTBS) protocol of rTMS over contralateral primary motor cortex will be applied.
  Interventions: Device: cTBS3

INTERVENTIONS:
Device: High-Frequency1 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% resting motor threshold (RMT), 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: ipsilateral primary motor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: High-Frequency1
Device: cTBS1 — rTMS intervention: 40 seconds of cTBS at 70% RMT, totaling 600 pulses.
  rTMS target: contralateral primary motor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: cTBS1
Device: High-Frequency2 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% RMT, 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: ipsilateral premotor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: High-Frequency2
Device: cTBS2 — rTMS intervention: 40 seconds of cTBS at 70% RMT, totaling 600 pulses.
  rTMS target: contralateral primary motor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: cTBS2
Device: High-Frequency3 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% RMT, 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: contralateral primary motor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: High-Frequency3
Device: cTBS3 — rTMS intervention: 40 seconds of cTBS at 70% RMT, totaling 600 pulses.
  rTMS target: contralateral primary motor cortex.
  Total rTMS sessions: once a day, 5 days per week, for 2 weeks, totaling 10 sessions.
  Additional treatment: inpatient conventional rehabilitation therapy, consisting of occupational and physical therapy for 30 minutes each, twice daily, for 2 weeks, as well as the routine pharmacotherapy based on the guidelines for management of patients with stroke.
  Arms: cTBS3

SUMMARY:
The objective of this study was to determine the effects of protocols of repetitive transcranial magnetic stimulation (rTMS) therapy based on the functional reserve of each hemiplegic stroke patient in subacute phase, compared to conventional low-frequency rTMS therapy on contralateral M1. Investigators hypothesized that the functional reserve of each hemiplegic stroke patient will be different, and therefore an appropriate simulating target for rTMS therapy is needed. In addition, this approach could be more effective compared to conventional protocols applied to stroke patients regardless of their severity, predicted mechanism of motor function recovery, or functional reserves.

DETAILED DESCRIPTION:
rTMS treatment for patients with stroke is traditionally based on interhemispheric interactions. The widely-used traditional rTMS treatment protocol involves inhibitory low-frequency or continuous theta burst stimulation (cTBS) applied over the contralesional hemisphere and excitatory high-frequency stimulation over the ipsilesional hemisphere. However, concerns have arisen regarding the effect of rTMS on motor recovery in stroke patients. Although still subject to debate, a possible reason for the diverse results of rTMS applied to stroke patients is the uniform application protocol to individuals with varying pathologies and functional reserves, aimed at enhancing recovery.

Therefore, this study was aimed to determine the effects of protocols of rTMS therapy based on the functional reserve of each hemiplegic stroke patient.

Based on screening evaluations (TMS-induced motor evoked potential (MEP), diffusion tensor imaging (DTI), MRI), investigators hypothesized that patients could be categorized into three groups: 1) preserved ipsilateral corticospinal tract, 2) preserved ipsilateral alternative corticospinal tract, and 3) no ipsilateral corticospinal tract preserved. For each group, investigators plan to randomly assign patients to experimental and control groups to demonstrate the efficacy of different rTMS protocols based on functional reserves compared to conventional inhibitory rTMS applied to the contralesional primary motor cortex.

ELIGIBILITY:
Inclusion Criteria:

1. hemiplegic stroke patients in the subacute phase (7 days to 3 months from the onset) who are currently hospitalized,
2. FMA score of the upper extremity ≤42,
3. adequate language and cognitive function to perform at least a 1-step obey-command,
4. pre-stroke functional level of modified Rankin Scale (mRS) ≤1,
5. aged ≥19 years old,
6. patients willing to sign the informed consent.

Exclusion Criteria:

1. those with contraindications to rTMS, such as epilepsy, implanted metal objects in the head, or a history of craniotomy,
2. those with progressive of hemodynamically unstable medical conditions,
3. those with coexisting neurological conditions, such as spinal cord injury or Parkinson's disease,
4. those with major psychiatric disorders, such as major depression, schizophrenia, or dementia,
5. those having contraindications to conduct an MRI study,
6. those who are pregnant or lactating ,
7. patients who have refused to participate in this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences of Fugl-Meyer Assessment score of Upper Extremity (FMA-UL) | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement for motor function of upper limb. Minimum: 0, Maximum: 66. Higher score means a better

SECONDARY OUTCOMES:
Differences of Fugl-Meyer Assessment score of Upper Extremity (FMA-UL) | From baseline T0 to During-intervention T1 (1 week)
  Measurement for motor function of upper limb. Minimum: 0, Maximum: 66. Higher score means a better
Differences of Fugl-Meyer Assessment score of Upper Extremity (FMA-UL) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for motor function of upper limb. Minimum: 0, Maximum: 66. Higher score means a better
Differences of Fugl-Meyer Assessment score (FMA) | From baseline T0 to During-intervention T1 (1 week)
  Measurement for motor function of all limbs. Minimum:0, Maximum: 100. Higher score means a better
Differences of Fugl-Meyer Assessment score (FMA) | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement for motor function of all limbs. Minimum:0, Maximum: 100. Higher score means a better
Differences of Fugl-Meyer Assessment score (FMA) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for motor function of all limbs. Minimum:0, Maximum: 100. Higher score means a better
Differences of Fugl-Meyer Assessment score of Lower Extremity (FMA-LL) | From baseline T0 to During-intervention T1 (1 week)
  Measurement for motor function of lower limb. Minimum:0, Maximum: 34. Higher score means a better
Differences of Fugl-Meyer Assessment score of Lower Extremity (FMA-LL) | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement for motor function of lower limb. Minimum:0, Maximum: 34. Higher score means a better
Differences of Fugl-Meyer Assessment score of Lower Extremity (FMA-LL) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for motor function of lower limb. Minimum:0, Maximum: 34. Higher score means a better
Differences of Box and block test | From baseline T0 to During-intervention T1 (1 week)
  Measurement for gross manual dexterity. Scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds.
Differences of Box and block test | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement for gross manual dexterity. Scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds.
Differences of Box and block test | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gross manual dexterity. Scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds.
Differences of Functional Ambulation Category (FAC) | From baseline T0 to During-intervention T1 (1 week)
  Measurement for gait function. Minimum: 0, Maximum: 5 Higher score means a better.
Differences of Functional Ambulation Category (FAC) | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement for gait function. Minimum: 0, Maximum: 5 Higher score means a better.
Differences of Functional Ambulation Category (FAC) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function. Minimum: 0, Maximum: 5. Higher score means a better.
Differences of Action Research Arm Test (ARAT) | From baseline T0 to During-intervention T1 (1 week)
  Measurement to assess upper extremity performance (coordination, dexterity and functioning).
  Minimum: 0, Maximum: 57. Higher score means a better.
Differences of Action Research Arm Test (ARAT) | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement to assess upper extremity performance (coordination, dexterity and functioning).
  Minimum: 0, Maximum: 57. Higher score means a better.
Differences of Action Research Arm Test (ARAT) | From baseline T0 to Follow-up T3 (2 months)
  Measurement to assess upper extremity performance (coordination, dexterity and functioning).
  Minimum: 0, Maximum: 57. Higher score means a better.
Differences of Jebsen-Taylor hand function test | From baseline T0 to During-intervention T1 (1 week)
  Measurement of fine and gross motor hand function using simulated activities of daily living.
  Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
Differences of Jebsen-Taylor hand function test | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement of fine and gross motor hand function using simulated activities of daily living.
  Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
Differences of Jebsen-Taylor hand function test | From baseline T0 to Follow-up T3 (2 months)
  Measurement of fine and gross motor hand function using simulated activities of daily living.
  Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
Differences of Hand grip strength test | From baseline T0 to During-intervention T1 (1 week)
  Measurement of muscular strength or the maximum force generated by forearm muscles, measured by Jamar hydraulic hand dynamometer.
Differences of Hand grip strength test | From baseline T0 to Post-intervention T2 (2 weeks)
  Measurement of muscular strength or the maximum force generated by forearm muscles, measured by Jamar hydraulic hand dynamometer.
Differences of Hand grip strength test | From baseline T0 to Follow-up T3 (2 months)
  Measurement of muscular strength or the maximum force generated by forearm muscles, measured by Jamar hydraulic hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Won Hyuk Chang, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HS, Kim DH, Seo HG, Im S, Yoo YJ, Kim NY, Lee J, Kim D, Park HY, Yoon MJ, Kim YS, Kim H, Chang WH. Efficacy of personalized rTMS to enhance upper limb function in subacute stroke patients: a protocol for a multi-center, randomized controlled study. Front Neurol. 2024 Jul 3;15:1427142. doi: 10.3389/fneur.2024.1427142. eCollection 2024. PMID 39022726